CLINICAL TRIAL: NCT03668717
Title: Survivorship and Outcomes of Robotic-Arm Assisted Medial Unicompartmental Knee Arthroplasty
Status: Active, not recruiting | Type: Observational
Sponsor: St. Helena Hospital Coon Joint Replacement Institute (Other)
Collaborators: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Other Study IDs: 004
Record Dates: First submitted 2016-09-28; First posted 2018-09-13 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis; medial; unicompartmental
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Robotic-arm assisted medical MCK implant — Robotic-arm assisted medical MCK implant system to replace the medial compartment of the knee.

SUMMARY:
The purpose of the study is to determine the survivorship of robotic-arm assisted MCK medial onlay Unicompartmental knee arthroplasty implants at two, five and tem year follow up.

DETAILED DESCRIPTION:
The purpose of the study is to determine the survivorship of robotic-arm assisted MCK medial onlay unicompartmental knee arthroplasty implants at two, five, and ten year follow up. Study participants will also be asked about their level of satisfaction with their knee function following their robotic-arm assisted Unicompartmental Arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* All patients over 21 years of age who underwent primary robotic-arm assisted unicompartmental arthroplasty and received a medial MCK onlay implant and are at least 24 months post-operative.
* Patient has signed an IRB approved Informed Consent Form or with IRB approved waiver of written consent, patient has verbally consented to study participations.
* Patient willing to comply with follow up.

Exclusion Criteria:

* Patient will be excluded from participation in the study if they are cognitively unable to answer questions related to their index procedure and health related quality of life forms.
* Patient had active infection
* Medial MCK onlay implants were implanted without bone cement
* Patients did not have sufficient bone stock to allow for insertion and fixation of components
* Patient did not have sufficient soft tissue integrity to allow for stability
* Patient had a neurological or muscular deformity that did not allow for control of the knee.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients over 21 years of age who required a primary robotic-arm assisted medial unicompartmental arthroplasty.
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2011-10; Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
% of patients with revisions | 10 year after surgery
  To determine the revision rate in this patient population

SECONDARY OUTCOMES:
% of patients with revisions | 2 years after surgery
  To determine the revision rate in this patient population

OTHER OUTCOMES:
% of patients with revisions | 5 years after surgery
  To determine the revision rate in this patient popluation

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Coon, MD, Principal Investigator — St. Helena Hospital Coon Joint Replacement Institute
Locations (1):
- St. Helena Hospital Coon Joint Replacement Institute, St. Helena, California, United States

IPD SHARING:
Plan to Share IPD: No